CLINICAL TRIAL: NCT01998438
Title: A Randomized Double-blinded Trial to Explore the Optimum Dose of Tranexamic Acid in Cardiopulmonary Bypass Cardiac Surgery
Brief Title: Prospective Trial of Tranexamic Acid in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hongwen Ji (Other)
Responsible Party: Sponsor-Investigator, Hongwen Ji, professor of medicine, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011GWH1
Record Dates: First submitted 2013-11-12; First posted 2013-11-28 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: tranexamic acid; cardiac surgery; cardiopulmonary bypass
MeSH Terms: interventions — Tranexamic Acid; Short Interspersed Nucleotide Elements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- small dose (Experimental): 10mg/kg tranexamic acid add in priming fluid, 10mg/kg single shot slowly when incision, followed by 2mg/(kg·h) infusion until the end of surgery
  Interventions: Drug: Tranexamic Acid
- medium dose (Experimental): 20mg/kg tranexamic acid add in priming fluid, 20mg/kg single shot slowly when incision, followed by 4mg/(kg·h) infusion until the end of surgery
  Interventions: Drug: Tranexamic Acid
- large dose (Experimental): 30mg/kg tranexamic acid add in priming fluid, 30mg/kg single shot slowly when incision, followed by 6mg/(kg·h) infusion until the end of surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — The loading doses were given in 15 minutes when incision.
  Other Names: SINE; Tranexamic Acid Injection; 120902

SUMMARY:
Tranexamic acid, an antifibrinolytic drug, is wildly used in cardiac surgeries to decrease perioperative bleeding and allogenic transfusion. But the optimum dose of tranexamic acid is still unknown. We use three different doses to find which is the optimum dose of tranexamic acid in cardiopulmonary bypass cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Noncyanotic congenital heart disease patients requiring cardiac surgeries under cardiopulmonary bypass
* Rheumatic or recessive valvular disease patients requiring valvular repair or replacement under cardiopulmonary bypass
* Coronary artery disease patients requiring coronary artery bypass graft under cardiopulmonary bypass

Exclusion Criteria:

* Non-primary and emergency cardiac surgery
* Disorder in coagulation function before surgery
* Anemia before surgery
* Definite liver and renal dysfunction
* History of stroke
* Pregnancy and lactation
* Disabled in spirit or law
* Fatal conditions such as cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 955 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongwen Ji, MD, Study Chair — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC; Haisong Lu, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Small Dose | Medium Dose | Large Dose
Started | 319 | 318 | 318
Completed | 319 | 318 | 318
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Small Dose | Medium Dose | Large Dose | Total
Number analyzed (Participants) | 319 | 318 | 318 | 955
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.9) | 53.2 (11.8) | 53.1 (11.6) | 53.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 138 | 138 | 413
  Male | 182 | 180 | 180 | 542

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Blood Loss
Time Frame: 24hrs postoperatively
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Small Dose | Medium Dose | Large Dose
Number analyzed (Participants) | 319 | 318 | 318
ml | 520 [350 to 690] | 490 [350 to 690] | 450 [324.5 to 620]

2. Secondary Outcome: Number of Participants Needs Allogenic Transfusion
Time Frame: on the 7th day postoperatively
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Rate of Reexploration for Bleeding
Time Frame: on the 7th day postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 days postoperative
Arm/Group | Small Dose | Medium Dose | Large Dose
Serious Adverse Events (participants affected / at risk) | 34/319 | 42/318 | 29/318
Other Adverse Events (participants affected / at risk) | 2/319 | 3/318 | 2/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Dose (N=319) | Medium Dose (N=318) | Large Dose (N=318)
renal dysfunction (Renal and urinary disorders) | 30 (30) | 40 (40) | 28 (28)
usage of IABP (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
cerebral embolism (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Small Dose (N=319) | Medium Dose (N=318) | Large Dose (N=318)
wound infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No